CLINICAL TRIAL: NCT03043742
Title: Prospective Controlled Trial of Intra-Myocardial Infusion of Bone Marrow Derived Autologous CD133+ Selected Cells During Trans-Myocardial Laser Revascularization (TMR) in Patients With Chronic Ischemic Heart Disease
Brief Title: Stem Cell Heart Injections During Laser Revascularization Surgery for Treatment of Chronic Ischemic Heart Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Sekela (Other)
Responsible Party: Sponsor-Investigator, Michael Sekela, Cardiothoracic Surgeon, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-1051
Record Dates: First submitted 2016-06-17; First posted 2017-02-06 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Chronic Ischemic Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I Open Label (Experimental): open label bone marrow derived autologous CD133+ selected stem cell application in patients receiving trans-myocardial laser revascularization to improve regional myocardial function as detailed below:
  Drug: CD133+ selected stem cells Dosage: Single injection of 0.1-0.2 ml around each laser channel Frequency: 10-20 channels Duration: Trans-Myocardial Revascularization
  Interventions: Drug: Bone Marrow Derived Autologous CD133+ Selected Cell Product

INTERVENTIONS:
Drug: Bone Marrow Derived Autologous CD133+ Selected Cell Product — Injection of bone marrow derived autologous CD133+ cell product into laser channels during Trans-Myocardial Revascularization
  Other Names: Stem cell

SUMMARY:
Assess the safety and effectiveness of stem cell application with regard to improvement in regional myocardial function in patients receiving Trans-Myocardial Laser Revascularization (TMR) and stem cells.

DETAILED DESCRIPTION:
Multiple case experiences and studies have been published reviewing clinical experiences with Carbon Dioxide Trans-Myocardial Laser Revascularization (TMR) and autologous bone marrow derived cell application. These experiences have demonstrated perfusion improvements, ejection fraction improvements and improvements in angina or heart failure symptoms. The investigators elected to examine the use of CD133 positive (CD133+) BM-derived stem cells because of their pluripotent nature and the fact that during the CD133 selection process inflammatory cells present in the bone marrow are being discarded. CD133+ is a recently discovered marker for more primitive bone marrow derived multipotent stem and endothelial progenitor cells and is of particular interest in studies directed to therapeutic angiogenesis, as these cells have been shown to differentiate into endothelial and myogenic cell lines. Multiple studies have utilized BM derived cells for myocardial regeneration. Patients who received CD133+ cells showed improved perfusion at injection sites of stem cells leading to a significant increase in volume of left ventricular ejection fraction, regional wall motion in the infarct zone, and a reduction in end systolic left ventricular volume.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two vessel coronary artery disease not amenable to direct revascularization
* Area of interest defined as part of free left ventricular vall with reduced contractility
* Demonstration of reduced perfusion in the area of interest (>30% of free wall)
* Global ejection fraction 30-45% with symptoms class >_ II on the NYHA scale
* Significant refractory angina defined as symptoms class >_ III that are refractory to maximal medical and anti-angina therapy
* Expected survival of at least two years

Exclusion Criteria:

* Any condition that prevents successful stem cell collection or application, e.g. systemic infection, puncture for stem cell collection impossible
* Any condition that may adversely affect bone marrow such as malignancy or prior irradiation to the pelvic bone
* Mitral valve insufficiency > moderate grade
* History of ventricular arrhythmias not controlled by medication and/or AICD
* Need for additional heart surgery (i.e. valve replacement)
* Emergency or salvage operation defined as within 48 hours of diagnosis
* Evidence of left ventricular thrombus
* Previous heart surgery within the last 6 months
* Increased Troponin T (> 3X ULN) in patients with unstable angina at time of intervention
* History of symptomatic carotid disease within the last 3 months prior to study intervention
* Ejection fraction < 30%
* End stage renal disease
* Untreatable cancer, current or within preceding 5 years
* Severe COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of Treatment-emergent serious adverse events (SAE) and adverse events | Assess from Procedure through 12 months
  Major adverse cardiac event and adverse events defined in the common toxicity criteria

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction compared to baseline | Assessed at baseline, 6 months, and 12 months
  Measured as a percentage by Echocardiography
Change in myocardial regional function compared to baseline | Assessed at baseline and 6 months
  Measured by nuclear scanning.
Change in myocardial regional viability compared to baseline | Assessed at baseline and 6 months
  Measured by nuclear scanning.
Change in distance walked compared to baseline | Assessed at baseline, 3 months, 6 months, and 12 months
  Measured in feet during a 6 minute walk test
Change in quality of life associated with heart failure compared to baseline | Assessed at baseline, 3 months, 6 months, and 12 months
  Measured using the Kansas City Cardiomyopathy Questionnaire.
Change in class of angina compared to baseline | Assessed at baseline, 3 months, 6 months, and 12 months.
  Measured using the Canadian Cardiovascular Society Grading Scale.
Change in class of heart failure compared to baseline | Assessed at baseline, 3 months, 6 months, and 12 months.
  Measured using the New York Heart Association Questionnaire
Change in regional left ventricular wall motion compared to baseline | Assessed at baseline, 6 months, and 12 months
  Measured using echocardiogram.
Change in quality of life associated with angina compared to baseline | Assessed at baseline, 3 months, 6 months, and 12 months
  Measured using the Seattle Angina Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sekela, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Healthcare, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
to be determined per principal investigator and statistician